CLINICAL TRIAL: NCT01756989
Title: ANGIOCOMB Antiangiogenic Therapy for Pediatric Patients With Diffuse Brain Stem and Thalamic Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Kuopio University Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Sanna-Maria Kivivuori, Sanna-Maria Kivivuori/Consultant in Pediatric Hematology and Oncology, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Angiocomb
Record Dates: First submitted 2011-05-18; First posted 2012-12-28 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Brainstem Glioma
MeSH Terms: interventions — Thalidomide; Etoposide; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide, etoposide, celecoxib (Experimental): Single arm study,phase II
  Interventions: Drug: Thalidomide, etoposide, celecoxib

INTERVENTIONS:
Drug: Thalidomide, etoposide, celecoxib — Thalidomide p.o. 1 mg/kg/day/1; the dose is gradually escalated, the maximum dose being 6 mg/kg/day. (The individual dose is set based on adverse effects.) Celecoxib p.o. 230 mg/m2/day/1-2, or in small children at 7 mg/kg/day in 1-2 doses.
  Etoposide p.o. the initial dosage 20 mg/m2/day; the dose is gradually escalated, the maxi 70 mg/m2/day.
  Other Names: vepesid (etoposide); celebra (celecoxib)

SUMMARY:
The purpose of this study is to determine whether initial local irradiation with topotecan and following oral antiangiogenic drugs, thalidomide, celecoxib and etoposide are effective in the treatment of pediatric diffuse brainstem tumor.

DETAILED DESCRIPTION:
All pediatric patients (aged 1-16 yrs) with newly diagnosed diffuse brain stem tumor or inoperable thalamic tumor which infiltrate brain stem from the pediatric oncology units in Denmark, Finland, Iceland, Norway and Sweden will be eligible. A possible tumor biopsy with histologic findings is not taken into account. The diagnosis is based on MRI. The patients are given a conventional local radiotherapy of 54 Gy, during which the patient also receives topotecan as radiosensitizer. Within four weeks after completed radiotherapy, the investigational drugs are started. If the family for some reason refuses radiotherapy, the investigational therapy may still be considered. The guardians and age-appropriate patients are asked for written informed consent. If the family is not willing to participate in the trial, the patient is treated according to the currently best available therapy (meaning RT without topotecan as palliative therapy). The family has the right to withdraw from the study, whenever they so wish.

Brain MRI at initial diagnosis, before the start of triple medication, and q 3 mo after initiation of triple medication, if not otherwise clinically indicated. In case it is decided to continue medication with progression in MRI, repeat MRIs are recommended every month. MRI should also be registered, if feasible, at the discontinuation of the medication.

The clinical follow-up, as well as MRI follow-up, on clinical indications will continue also after discontinuation of therapy.

PET-CT and/or MRI spectroscopy should be considered at diagnosis and at 3 mo after the start of triple medication.

ELIGIBILITY:
Inclusion Criteria:

-pediatric diffuse brainstem tumor

Exclusion Criteria:

* wish of the family
* need for strong painrelievers
* decreased level of consciousness
* inability to swallow.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2005-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Survival | up to five years
  Primary outcome measure is survival in months.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna-Maria Kivivuori, md, Study Chair — Helsinki University Central Hospital
Locations (1):
- Div of Hem/Onc and SCT, Children's Hospital, HUCH, Helsinki, Finland